CLINICAL TRIAL: NCT00607503
Title: A Pilot Study to Evaluate the Safety of Terbutaline in Children With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DirecNet 010; HD041919-01; HD041915-01; HD041890; HD041918-01; HD041908-01; HD041906-01; M01RR000069 (NIH); RR00059; RR 06022; RR00070-41.
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Terbutaline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Terbutaline

INTERVENTIONS:
Drug: Terbutaline — Each subject will be treated with terbutaline for 21-28 days following the initiation of treatment during the CRC admission.
  Subjects weighing between 25 and 45 kg will be treated with a nightly oral dose of 2.5 mg and subjects who weigh more than 45 kg will be treated with 3.75 mg.
  The standard 2.5 mg terbutaline tablets available in a pharmacy will be used in the study, with subjects taking either 1 or 1.5 tablets nightly.
  Other Names: Brethine

SUMMARY:
The purpose of the study is to gain experience with the use of terbutaline in children with T1D and to determine that there is not a frequent serious, unexpected, uncontrollable effect on short-term glycemic control. Some information also will be obtained with regard to whether terbutaline, in the dosing being used in the study, is sufficiently well tolerated to expect that adherence will be satisfactory in a large randomized trial. In addition, this pilot study will provide data on the accuracy of a continuous glucose monitor during terbutaline use to verify that the drug does not impact on sensor function.

DETAILED DESCRIPTION:
Approximately 10 children will be recruited from five centers in the United States to participate in this study. The data collected in this pilot study will be used to determine whether to proceed to a randomized trial using the dose of terbutaline being used in the pilot study or the need for additional pilot testing with a lower dose of terbutaline.

Beginning the Study

When a chid enters the study, the following will be done:

1. After eligibility is determined, informed consent and assent are obtained from the parent/guardian and subject.
2. An unblinded CGM will be used and blood ketones will be checked each morning by the subject for at least one week. Subjects may be asked to wear an Actiwatch monitor each night.
3. Terbutaline will be initiated during a CRC admission and continued following the CRC stay for 21-28 days.

   • Subjects weighing between 25 and 45 kg will be treated with a nightly oral dose of 2.5 mg and subjects who weigh more than 45 kg will be treated with 3.75 mg.
4. The CRC admission will last approximately 18-20 hours and include the following:

   * Monitoring of effects of terbutaline by measurement of heart rate, blood pressure, blood and interstitial glucose, lactate, ketones, NEFA, B-OH butyrate
   * Assessment of the accuracy of the CGM by comparing sensor glucose values to blood glucose values
5. The outpatient phase will last 21-28 days and include the following:

   * Nightly use of terbutaline as described above
   * Use of an unblinded CGM on a daily basis to monitor the glucose levels
   * Subjects may be asked to wear the Actiwatch monitor overnight
   * Measurement of blood ketones each morning
   * Phone calls to each subject on the first outpatient day of terbutaline use and then approximately every 3 days (twice a week) until the end of the subject's follow up.
6. Second CRC admission to mirror the first admission between 21 and 28 days after initiation of terbutaline
7. Follow up for 1-2 weeks after discontinuation of terbutaline until glucose control is back to prestudy level.

Procedures at home after hospital stay

1. Terbutaline will be taken orally each day prior to bedtime.
2. Each subject will continue to use a CGM, with instructions to use it as close to 24/7 as possible.
3. Prior to each phone call, the subject will be instructed to download the CGM and either email or fax the file to the clinic so that the glucose data can be reviewed during the phone contacts.
4. Each subject will be provided with an HGM and test strips. The HGM will be used for calibration of the CGM and to confirm high and low values on the CGM prior to acting on them. It will be downloaded at the end-of-study CRC admission. The subject will be asked to measure blood ketones each morning using the meter and strips that will be provided.
5. Each subject may be asked to wear an Actiwatch each night to measure movement while the subject is sleeping.
6. Phone calls to each subject will be made after the first outpatient day of terbutaline use and then approximately every 3 days (twice a week) until the end of the subject's follow up plus an about 7 days after terbutaline is discontinued.
7. Prior to the end-of-study CRC admission, follow-up visits can occur at any time at the discretion of the investigator.

End of study admission

The end-of study CRC admission will occur after 21-28 days of the outpatient phase.The protocol will be identical to the protocol for the first CRC admission. The dinner and breakfast meals will be identical to the meals given during the first admission.

The sensors will be removed prior to discharge, unless the investigator decides it would be beneficial to continue a CGM for 1-2 weeks to assist in the maintenance of glucose control after terbutaline has been stopped.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
* Age 12.0 years to less than 18.0 years
* HbA1c <8.0%
* Use of basal: bolus insulin therapy with either an insulin pump or glargine with MDI of a short-acting insulin for at least 6 months (approximately 5 pump and 5 MDI users will be enrolled)
* Availability of home computer to download the CGM
* For females: not currently pregnant, negative pregnancy test, and not intending to become pregnant during the next 3 months
* Parent/guardian and subject understand the study protocol and agree to comply with it
* Informed Consent Form signed by the parent/guardian and Child Assent Form signed by the subject if required by IRB

Exclusion Criteria:

* Severe hypoglycemic event (seizure or coma) or diabetic ketoacidosis in the past 6 months
* Cardiac disease, including prolonged QT interval on EKG or pathologic arrhythmia
* An EKG will be done either prior to the CRC admission or during the CRC admission prior to the first dose of terbutaline
* Treatment for hypertension or blood pressure exceeding the 90th percentile for age and height
* Current treatment for a seizure disorder
* Asthma if treated with systemic or inhaled corticosteroids in the last 6 months or with a beta adrenergic agonist more than once a month
* Cystic fibrosis
* Use of MAO inhibitors, tricyclic antidepressants, or beta blockers
* Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
* Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian).
* Medical condition that in the judgment of the investigator might interfere with the completion of the protocol

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety of bedtime administration of the epinephrine simulating β2 adrenergic agonist terbutaline to reduce the incidence of nocturnal hypoglycemia without compromising glycemic control in youth with type 1 diabetes (T1D). | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Roy W Beck, MD, PhD, Study Director — Jaeb Center for Health Research
Locations (6):
- United States (6):
  - Division of Pediatric Endocrinology and Diabetes, Stanford University, Stanford, California
  - Department of Pediatrics, Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jaeb Center for Health Research, Tampa, Florida
  - Department of Pediatrics, University of Iowa Carver College of Medicine, Iowa City, Iowa
  - Washington University, St Louis, Missouri